CLINICAL TRIAL: NCT00853463
Title: Multi-centered Discharge Alert to Prevent DVT and PE at Hospital Discharge
Brief Title: Discharge ALERT: Quality Improvement Initiative
Acronym: Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Samuel Goldhaber, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-P-001083
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Prophylaxis; Venous Thromboembolism; Prevention
Keywords: Pulmonary Embolism; Deep Vein Thrombosis; Prophylaxis; Venous thromboembolism; Prevention; Medical patients
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism | interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Alert (No Intervention): The responsible physician of a patient randomized to the control arm will not be contacted regarding the increased VTE risk of the patient.
- Alert (Other): The responsible physician will be notified that: 1) his or her patient is at high risk for VTE and 2) VTE prophylaxis should be considered in the Discharge orders
  Interventions: Behavioral: Alert

INTERVENTIONS:
Behavioral: Alert — The responsible physician will be notified that: 1) his or her patient is at high risk for VTE and 2) VTE prophylaxis should be considered in the Discharge orders
  Other Names: "Alert"
  Arms: Alert

SUMMARY:
Brigham and Women's Hospital will coordinate a Quality Improvement Initiative at other hospitals that focuses on whether physician notification prior to discharge of high risk VTE patients will reduce the incidence of VTE after hospital discharge.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION AND RATIONALE FOR THE STUDY

Venous thromboembolism (VTE) is often avoidable in hospitalized patients because proven prevention strategies have been established for patients at risk (1). North American and European prophylaxis guidelines have been widely disseminated. However, despite focus on strategies for the prevention of VTE in hospitalized patients at the time of admission to the hospital, there has been little focus on prevention of VTE at the time of discharge from the hospital (2,3).

At Brigham and Women's Hospital, we undertook a previous Quality Improvement Initiative (BWH protocol # 2000P000328) aimed at increasing the frequency of VTE prophylaxis in high risk patients. This novel strategy required: 1) devising a risk score that reliably and quickly identified patients at high risk of VTE, and 2) randomizing high-risk patients without prophylaxis into an intervention group or control group. The intervention group's physicians received a single electronic, computerized alert explaining that the patient was at high risk, was not receiving prophylaxis, and suggesting that prophylaxis be ordered from a template of available pharmacological and mechanical options. In contrast, the control group's physicians received no alert (4).

Each of 8 common risk factors was weighted according to a point scale. To be labeled as "high-risk" for VTE, the point score must equal or exceed 4 points.

There were 2,506 patients in the Quality Improvement Initiative: 1,255 in the intervention group and 1,251 in the control group. The incidence of symptomatic VTE at 90 days was high: 8.2% in the control group and 4.9% in the intervention group (4).

Currently, an investigator initiated Quality Improvement Initiative (BWH protocol # 2005-P-002527) of human alerts rather than electronic, computerized alerts, has been undertaken in high risk patients not receiving prophylaxis. Enrollment of 2,500 patients at 25 centers located throughout the United States was completed in November 2007 with a follow-up rate that exceeded 99%. Analysis of the data is currently being conducted.

Limited research focus has been placed on high-risk VTE subjects in the community, outside of the hospital setting. Since most VTE prophylaxis has focused upon protection of high-risk patients at the time of hospital admission, there is a need to focus on VTE prophylaxis within 48 hours of hospital discharge. It is clear that as preparations are being made for hospital discharge, many patients remain at high risk for DVT and acute pulmonary embolism. After discharge, some patients will have an even higher risk than during hospitalization because of prolonged immobilization and bed rest at home (5).

The Discharge Alert Quality Improvement Initiative will determine whether alerting physicians about the importance of continued VTE prophylaxis just prior to the time of planned hospital discharge will lower the incidence of outpatient VTE. This new strategy is unproven and might not be effective, but this Quality Improvement Initiative should provide a definitive answer.

We will also implement as part of our Discharge Alert Trial an in-hospital Quality Improvement Initiative of intensive patient education at Brigham and Women's Hospital to improve patient adherence to physician-ordered pharmacological venous thromboembolism (VTE) prophylaxis. We hypothesize that after implementation of this education program, fewer patients will decline physician-ordered doses of enoxaparin or unfractionated heparin (UFH) compared with a recent cohort of patients at risk for VTE who did not receive specialized education about VTE.

METHODOLOGY

Identification of Patients at Risk for Venous Thromboembolism (VTE)

Hospitalized patients awaiting planned discharge within 48 hours will be evaluated with a previously validated (BWH protocol # 2000P000328) VTE risk profile. The VTE risk profile will be computed for each patient awaiting discharge using 8 common risk factors. Each risk factor is weighted according to a point score. To be labeled as "high risk" for VTE, the point score must equal or exceed 4 points.

Minor (Low) Risk Factors (1 POINT each):

* Advanced Age (> 70 years of age)
* Obesity (BMI > 29, or the presence of the word "obesity" in admission exam notes)
* Bed rest / Immobility (not related to surgery)
* Female Hormone Replacement Therapy or Oral Contraceptives

Intermediate Risk Factor (2 POINTS each):

* Major Surgery (> 60 minutes, during this admission)

Major (High) Risk Factors (3 POINTS each):

* Cancer (active)
* Prior VTE
* Hypercoagulability

Screening for Venous Thromboembolism Prophylaxis

If the cumulative VTE risk score is at least 4, orders are reviewed to detect ongoing mechanical or pharmacological prophylactic measures. Mechanical prophylactic measures include graduated compression stockings and intermittent pneumatic compression devices. Pharmacological prophylactic measures include unfractionated heparin, enoxaparin, dalteparin, fondaparinux, tinzaparin, and warfarin.

At Brigham and Women's Hospital, we will also identify all new orders for pharmacological VTE prophylaxis with enoxaparin and UFH using the BWH computerized order entry system as part of an additional component of the Quality Improvement Initiative. For this component of the Quality Improvement Initiative, eligibility is defined as having a DVT Risk Score of 3 or higher and having electronically entered physician's orders for appropriate pharmacologic VTE thromboprophylaxis.

Quality Improvement Intervention

The intervention will take place within 48 hours of planned hospital discharge. If randomized to the alert, the responsible physician will be notified that: 1) his or her patient is at high risk for VTE, and 2) VTE prophylaxis should be considered in the Discharge orders. If randomized to no alert (control patients), the responsible physician will not be contacted.

At Brigham and Women's Hospital, we will also provide 500 eligible patients in a prospective cohort with one-on-one education using a scripted dialog to describe the rationale and importance of pharmacological VTE prophylaxis.

Prophylaxis Guidelines at Discharge

"Consider Venous Thromboembolism prophylaxis at the time of hospital discharge in patients with congestive heart failure or respiratory disease or prolonged immobility."

"For those without contraindication, consider pharmacological prophylaxis with low-molecular weight heparin, unfractionated heparin, or fondaparinux."

"For those at high risk of bleeding, consider mechanical prophylaxis with intermittent pneumatic compression devices or graduated compression stockings."

Follow Up

A 90-day follow-up will be performed for all study patients. If patient outcomes cannot be determined by medical record review alone, then study representatives may contact the subject's Primary Care Physician (PCP) for necessary information. IRB approval must be obtained at each participating hospital prior to any contact with subjects' PCPs.

Data Collection and Study Endpoints

The primary endpoint is clinically diagnosed DVT or PE at 90 days. Safety endpoints include total mortality and hemorrhagic events at 90 and 30 days, respectively. These are the same endpoints utilized in our prior Quality Improvement Initiative (BWH protocol # 2000P000328).

Hemorrhagic events will be classified according to the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO) trial criteria. Bleeding events will be classified as severe or life-threatening if they are intracerebral or if they result in substantial hemodynamic compromise requiring treatment. Moderate bleeding is defined by the need for transfusion. Minor events refer to bleeding not requiring transfusion or causing hemodynamic compromise. We will report rates of "major bleeding" which will be defined as GUSTO severe/life-threatening or moderate bleeding.

For the additional component of the Quality Improvement Initiative at Brigham and Women's Hospital, we will also assess improvement of medication adherence with enoxaparin and UFH following an intensive and individualized patient education program compared with our recently completed cohort study in which no uniform education program was targeted at VTE prophylaxis.

Statistical Analysis

The initial sample size (power 80%, two-sided alpha 5%) has been calculated at 2,500 patients based on an estimated 7% rate of the primary end point in the control group, and an odds ratio of 0.59 for the primary endpoint in intervention group patients. This yields a sample size requirement of 2,138 patients, plus an estimated 362 patients who will withdraw from the study.

We will use Wilcoxon rank-sum tests for comparisons in the distributions of continuous variables between groups, and chi-square tests or Fisher's exact test for comparisons of categorical variables. The primary analysis is the difference in the Kaplan-Meier estimator for freedom from VTE at day 90 between intervention and control patients. The log-rank test will estimate the cumulative probability of the primary endpoint in the intervention and control groups. We will use the proportional-hazards model for estimation of the relative hazard of clinical endpoints associated with the physician alert. All p-values reported are two-sided.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Planned discharge within 48 hours
* Cumulative VTE risk score at least 4
* Patients from Medical Services

Exclusion Criteria:

* VTE risk score <4
* Patients <18 years of age
* Full anticoagulation therapy planned upon discharge, i.e., atrial fibrillation, mechanical heart valve, venous thromboembolism treatment, etc.
* Patient is admitted to a non-medical service, i.e., surgical service, orthopedics, obstetrics/gynecology, neurology, psychiatry, or other non-medical service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2515 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Clinically diagnosed DVT and/or PE | 90 days after discharge

SECONDARY OUTCOMES:
Mortality | 30 and 90 days
Hemorrhagic events | 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (22):
- United States (22):
  - Long Beach VA Healthcare System, Long Beach, California
  - UC Irvine, Orange, California
  - UC Davis, Sacramento, California
  - Denver VA Medical Center, Denver, Colorado
  - William Backus Hospital, Norwich, Connecticut
  - Medstar Research Frankin Square Hospital, Baltimore, Maryland
  - Washington County Hospital, Hagerstown, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - North Shore Medical Center, Salem, Massachusetts
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - University of Missouri- Columbia, Columbia, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Lovelace Medical Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - North Shore University Hospital, Manhasset, New York
  - Duke University Medical Center, Durham, North Carolina
  - Indiana Regional Medical Center, Indiana, Pennsylvania
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - Washington Hospital, Washington, Pennsylvania
  - Presbyterian Hospital Texas Health, Dallas, Texas
  - University of Utah Hospital Medical Center, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah

REFERENCES:
- [Background] Goldhaber SZ, Turpie AG. Prevention of venous thromboembolism among hospitalized medical patients. Circulation. 2005 Jan 4;111(1):e1-3. doi: 10.1161/01.CIR.0000150393.51958.54. No abstract available. PMID 15630031
- [Background] Goldhaber SZ, Dunn K, MacDougall RC. New onset of venous thromboembolism among hospitalized patients at Brigham and Women's Hospital is caused more often by prophylaxis failure than by withholding treatment. Chest. 2000 Dec;118(6):1680-4. doi: 10.1378/chest.118.6.1680. PMID 11115458
- [Background] Goldhaber SZ, Tapson VF; DVT FREE Steering Committee. A prospective registry of 5,451 patients with ultrasound-confirmed deep vein thrombosis. Am J Cardiol. 2004 Jan 15;93(2):259-62. doi: 10.1016/j.amjcard.2003.09.057. PMID 14715365
- [Background] Kucher N, Koo S, Quiroz R, Cooper JM, Paterno MD, Soukonnikov B, Goldhaber SZ. Electronic alerts to prevent venous thromboembolism among hospitalized patients. N Engl J Med. 2005 Mar 10;352(10):969-77. doi: 10.1056/NEJMoa041533. PMID 15758007
- [Background] Spencer FA, Lessard D, Emery C, Reed G, Goldberg RJ. Venous thromboembolism in the outpatient setting. Arch Intern Med. 2007 Jul 23;167(14):1471-5. doi: 10.1001/archinte.167.14.1471. PMID 17646600